CLINICAL TRIAL: NCT01169415
Title: Effects of Dexamethasone Tapering Schedules on Functional Capacity and Neurocognition in Patients With Newly Diagnosed Glioblastoma Multiforme
Brief Title: Effects of Steroid Tapering on Functional Capacity and Neurocognition
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding not obtained
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00024406
Record Dates: First submitted 2010-06-25; First posted 2010-07-26 (Estimated); Last update posted 2014-05-19 (Estimated); Status verified 2014-05

CONDITIONS: Glioblastoma Multiforme
Keywords: Randomized; Dexamethasone; Abbreviated; Protracted; Post-operatively
MeSH Terms: conditions — Glioblastoma | interventions — dexamethasone acetate; Calcium Dobesilate; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Protracted (30 days), Dexamethasone (Experimental): Participants will receive a protracted course (30 days) of dexamethasone after surgery.
  Interventions: Drug: Dexamethasone acetate
- Abbreviated (14 days), dexamethasone (Experimental): Participants will receive an abbreviated (14 days) course of dexamethasone after surgery.
  Interventions: Drug: Dexamethasone

INTERVENTIONS:
Drug: Dexamethasone acetate — Participants will receive a protracted (30 days) course of dexamethasone after surgery.
  Other Names: Decadron
  Arms: Protracted (30 days), Dexamethasone
Drug: Dexamethasone — Participants will receive a protracted (14 days) course of dexamethasone after surgery.
  Other Names: Decadron
  Arms: Abbreviated (14 days), dexamethasone

SUMMARY:
Purpose and Objective:

1. To compare the effects of either an abbreviated or protracted taper of dexamethasone on functional capacity in newly diagnosed glioblastoma multiforme (GBM) patients.
2. To compare neurocognitive function in newly diagnosed GBM patients receiving either an abbreviated or protracted taper of dexamethasone.
3. To compare skeletal muscle strength in newly diagnosed GBM patients receiving either an abbreviated or protracted taper of dexamethasone.
4. To examine the association between functional capacity and neurocognitive function and patient-reported measures (i.e. quality of life, fatigue, etc.) in newly diagnosed GBM patient on either an abbreviated or protracted taper of dexamethasone.
5. To examine the association between functional capacity and neurocognitive function and body composition measures (body-mass index, etc.) in newly diagnosed GBM patient on either an abbreviated or protracted taper of dexamethasone.
6. To examine the association between functional capacity and neurocognitive function and biochemical metabolic measurements in newly diagnosed GBM patient on either an abbreviated or protracted taper of dexamethasone.

All study endpoints will be assessed at three timepoints as follows: (1) initial assessment after surgery in the hospital, (2) second assessment at initial clinical visit at the Preston Robert Tisch Brain Tumor Center (PRT-BTC) at Duke, approximately 1 week post-operatively, and (3) third assessment at second clinical visit in the PRT-BTC at Duke, approximately 10 weeks post-operatively and after completion of radiotherapy. An additional fourth assessment will be obtained at 4 weeks post-operatively if the subject is undergoing radiotherapy here at Duke.

DETAILED DESCRIPTION:
The proposed study is a randomized controlled trial. After obtaining written informed consent, all participants will be randomized to either an abbreviated (14 days) or protracted (30 days) course of dexamethasone post-operatively.

ELIGIBILITY:
Inclusion Criteria:

1. written informed consent prior to beginning specific protocol procedures,
2. histologically proven GBM,
3. status-post gross total resection or subtotal resection as indicated by < 2 cm of residual enhancing disease (subjects with unresectable, multifocal, and /or bulky disease will be excluded),
4. >18 years and <70 years of age,
5. Karnofsky performance index >70%,
6. no documented cardiac, neurodegenerative, neuromuscular, or pulmonary disease,
7. no contraindications to a 6-minute walk test,
8. no contraindications to neurocognitive testing,
9. primary treating physician approval, and
10. no complications operatively or postoperatively that requires modification of dexamethasone dosing.
11. receiving dexamethasone as standard of care.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-06; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Functional Capacity (6-minute walk test) | 10 weeks
  The exercise test is designed to determine how far you can walk in six minutes. This test will take place at the PRT-BTC at Duke University Medical Center and/or Duke University Medical Center inpatient unit on 4100 or 4300 with appropriate medical supervision.

SECONDARY OUTCOMES:
Neurocognitive Function | 10 weeks
  A computerized neurocognitive test battery called CNS Vital Signs® including verbal memory test, visual memory test, finger tapping test, symbol digit coding, Stroop test, shifting attention test, continuous performance test.
Skeletal Muscle Strength | 10 weeks
  Isokinetic muscle strength for bilateral grip and bilateral quadriceps.
Patient-Reported Outcomes (PROs) | 10 weeks
  Assessed by standardized and validated questionnaires including: Depression (Beck Depression Inventory); Quality of Life (Functional Assessment of Cancer Therapy-Brain); Fatigue (Functional Assessment of Cancer Therapy-Fatigue); Cognition (Functional Assessment of Cancer Therapy-Cognition), Symptomalogy Index (Phone Questionnarie/Survery), Computerized Battery from CNS Vital Signs (Medical Outcomes Survey, Epworth Sleepiness Scale, Pittsburgh Sleep Quality Index, Zung Self-Rating Depression Scale).
Body composition | 10 weeks
  Body-mass index, weight, height, and circumference of the abdomen, hips, and quadriceps.
Biochemical metabolic measurements | 10 weeks
  Hematocrit (%), albumin (g/mL), fasting blood glucose (mg/dL), fasting insulin (micro IU/mL), insulin like growth facto binding protein 1 (IGFBP-1) (ng/mL), cystatin C (mg/dL), and retinol binding protein 4 (RBP-4).

CONTACTS AND LOCATIONS:
Overall Officials: Katherine B Peters, MD, PhD, Principal Investigator — Duke Health